CLINICAL TRIAL: NCT01934959
Title: A Prospective Multicenter Randomized Controlled Trial on Probiotics in Preventing Hirschsprung's Disease Associated Entercolitis
Brief Title: A Trial on Probiotics in Preventing Hirschsprung's Disease Associated Entercolitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jiexiong Feng, Chief of Pediatric Surgery, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Tongji
Record Dates: First submitted 2013-08-21; First posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Probiotics; Hirschsprung's Disease Associated Enterocolitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probiotics (Experimental)
  Interventions: Drug: Bifico

INTERVENTIONS:
Drug: Bifico

SUMMARY:
Enterocolitis(EC) is the most common and serious postoperative complication of Hirschsprung's disease(HD) with high morbidity and mortality. Probiotics are live microbes that, when administered in adequate amounts, confer health benefit to the host.Based on this previous knowledge on the beneficial effects of probiotics during pro-inflammatory conditions of the gastrointestinal tract, investigators hypothesized that oral probiotics could decrease the incidence and severity of Hirschsprung's disease associated enterocolitis(HAEC).Investigators conducted a prospective, multicenter, randomized and controlled trial to assess whether oral probiotics could decrease the incidence and severity of Hirschsprung's disease associated enterocolitis(HAEC).

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria consists of all patients suffering from HD at an age of less than 13 years old, and HD is confirmed by postoperative pathological examination, barium enema and anorectal manometry.

Exclusion Criteria:

* Age> 13 years old
* Patients are complicated with mental, neurological disorders (such as hypoxic-ischemic encephalopathy, epilepsy and dementia) or can not thrive.
* Patients are complicated with congenital gastrointestinal malformations (such as anal stenosis, intestinal atresia stenosis), metabolic and endocrine diseases caused by organic constipation and functional constipation in children.
* Children are complicated with liver, kidney dysfunction, blood disorders, immune deficiency diseases and significant ECG abnormalities.
* Children have taken oral antibiotics, microecological modulator, yogurt, other gastrointestinal motility drugs which can affect the gut flora.
* Drug allergies, or allergic diseases..
* Poor compliance with oral probiotics treatment.

Ages: 1 Month to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Probiotics Prevent Hirschsprung's Disease Associated Entercolitis | two years

REFERENCES:
- [Derived] Wang X, Li Z, Xu Z, Wang Z, Feng J. Probiotics prevent Hirschsprung's disease-associated enterocolitis: a prospective multicenter randomized controlled trial. Int J Colorectal Dis. 2015 Jan;30(1):105-10. doi: 10.1007/s00384-014-2054-0. Epub 2014 Nov 5. PMID 25370155